CLINICAL TRIAL: NCT05263401
Title: 3-hydroxybutyrate as a Meal Primer in Patients With Type 2 Diabetes
Brief Title: Keto Drinks as a Meal Primer in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1-10-72-282-20
Record Dates: First submitted 2021-12-14; First posted 2022-03-02 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2021-12

CONDITIONS: Type 2 Diabetes; Ketoses, Metabolic
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Ketosis | interventions — 3-Hydroxybutyric Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ketone salt (Experimental): Na-D/L-3-hydroxybutyrate dissolved in tap water.
  Interventions: Dietary Supplement: 3-hydroxybutyrate
- Ketone ester (Experimental): (R)-3-Hydroxybutyl (R)-3-hydroxybutyrate
  Interventions: Dietary Supplement: 3-hydroxybutyrate
- Placebo (Placebo Comparator): Tap water
  Interventions: Dietary Supplement: 3-hydroxybutyrate

INTERVENTIONS:
Dietary Supplement: 3-hydroxybutyrate — Orally administered pre-meal drinks.

SUMMARY:
The main objective of this clinical trial is to study the effects of orally administered ketone drinks containing the ketone body, 3-hydroxybutyrate (3-OHB), just before a meal in patients with type 2 diabetes. Moreover the investigators will compare the effects of two different ketone drinks.

The hypothesis is:

3-OHB as a pre-meal may:

* Lower postprandial blood glucose and lipids.
* Mediate release of intestinal hormones and affect gastric emptying.
* Affect appetite and other subjective measures related to food intake.

The effects of 3-OHB as a pre-meal will be investigated by blood samples, isotopic tracers examinations, paracetamol test, questionnaires and meal test.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes diagnosis, metformin treated or dietary treated
* HbA1C < 80 mmol/mol
* 25 < BMI < 35
* Written consent

Exclusion Criteria:

* Severe comorbidity
* Treatment with insulin, GLP-1 analogues, SGLT-2-inhibitors or sulfonylureas
* Specific diets, e.g. ketogenic diet
* PI finds the patient not fit (e.g. mental illness, too nervous, unacceptable screening blood tests or other)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Postprandial P-glucose | 3 hours
  Incremental area under the curve (iAUC) for P-glucose.

SECONDARY OUTCOMES:
Postprandial free fatty acids (FFA) | 3 hours
  Blood samples
Differences in circulating concentrations of 3-hydroxybutyrate | 3,5 hours
  Blood samples
Lipolysis rate | 3 hours
  Measures of palmitate flux (palmitate tracer)
Glucose kinetics | 3 hours
  Glucose tracer examinations
Gastric emptying | 3 hours
  Paracetamol test
Differences in hunger/satiety | 4 hours
  Questionnaire for quantifying hunger/satiety on a VAS scale from 1-10
Differences in actual hunger | 30 minutes
  Ad libitum meal test
Differences in circulating concentrations of insulin | 3,5 hours
  Blood samples
Differences in circulating concentrations of glucagon | 3,5 hours
  Blood samples
Differences in circulating concentrations of c-peptide | 3,5 hours
  Blood samples
Differences in circulating concentrations of Glucagon-like peptide-1 (GLP-1) | 3,5 hours
  Blood samples
Differences in circulating concentrations of Gastric inhibitory polypeptide (GIP) | 3,5 hours
  Blood samples
Differences in circulating concentrations of ghrelin | 3,5 hours
  Blood samples
Differences in circulating concentrations of cholecystokinin | 3,5 hours
  Blood samples
Differences in circulating concentrations of gastrin | 3,5 hours
  Blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Niels Møller, Professor, Study Director — Aarhus University Hospital
Locations (1):
- Medical research laboratory, Department of endocrinology, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bangshaab M, Bengtsen MB, Smedegaard S, Sondergaard E, Moller N, Svart MV, Rittig N. Ketone supplementation dose-dependently lowers postprandial blood glucose, lipid and ghrelin levels in individuals with type 2 diabetes: a randomised crossover study. Diabetologia. 2025 Nov 28. doi: 10.1007/s00125-025-06614-0. Online ahead of print. PMID 41315088